CLINICAL TRIAL: NCT03984357
Title: Induction, Concurrent and Adjuvant Nivolumab Combined With Induction Chemotherapy Followed by Radiotherapy Alone in Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase 2, Multi-center, Single-arm Clinical Trial
Brief Title: Nivolumab Combined With Chemoradiotherapy Sparing Concurrent Cisplatin in Nasopharyngeal Carcinoma
Acronym: PLATINUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jun Ma, MD, Principal Investigator, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7GC
Record Dates: First submitted 2019-06-07; First posted 2019-06-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: PD-1 blockade; immune checkpoint inhibitor; induction chemotherapy; radiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Immune Checkpoint Inhibitors; Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD-1 blocking antibody combined with IC+IMRT (Experimental): All participants will receive induction chemotherapy (IC; every 3 weeks × 3 cycles; gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1) followed by intensity-modulated radiotherapy (IMRT; 70 Gy, 33 fractions, 5 fractions/week, 1 fraction/day) alone. PD-1 blocking antibody (360 mg per cycle) will start on day 1 of the first cycle IC and continue every 3 weeks for 6 cycles till the end of IMRT, involving the whole-course of IC + IMRT alone. The first and last 3 cycles of PD-1 blocking antibody are administrated concurrently with IC and IMRT, respectively. After 4 weeks of the completion of IMRT, adjuvant PD-1 blocking antibody (480 mg per cycle) will begin every 4 weeks for 6 cycles.
  Interventions: Drug: PD-1 blocking antibody; Drug: Gemcitabine; Drug: Cisplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: PD-1 blocking antibody — 1. Whole-course concurrent PD-1 blocking antibody: every 3 weeks × 6 cycles; 360 mg, day 1; start on day 1 of the first cycle IC and continue every 3 weeks for 6 cycles till the end of IMRT, involving the whole-course of IC + IMRT alone.
  2. Adjuvant PD-1 blocking antibody: every 4 weeks × 6 cycles; 480 mg, day 1
  Other Names: PD-1 blockade
Drug: Gemcitabine — Gemcitabine as induction chemotherapy, 1000 mg/m2 day 1, 8 per cycle, every 3 weeks for 3 cycles
  Other Names: GEM
Drug: Cisplatin — Cisplatin as induction chemotherapy, 80 mg/m2 day 1 per cycle, every 3 weeks for 3 cycles
  Other Names: DDP
Radiation: Intensity-modulated radiotherapy — Definitive IMRT of 70 Gy, 33 fractions, 5 fractions/week, 1 fraction/day
  Other Names: IMRT

SUMMARY:
This is a phase 2, single-arm, multicenter clinical trial, with the purpose to evaluate the therapeutic efficacy, safety, and tolerability of PD-1 Blockade nivolumab combined with a deintensified chemoradiotherapy by sparing concurrent cisplatin from the standard induction chemotherapy plus concurrent chemoradiotherapy in high-risk locoregionally advanced nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This phase 2, single-arm, multicenter clinical trial plans to enroll 152 patients with newly-diagnosed, pathologically-proven, untreated locoregionally advanced nasopharyngeal carcinoma (LANPC) at high-risk of distant metastasis (T4N1M0 or T1-4N2-3M0, according to American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC] 8th edition clinical staging system). Patients will receive 3 cycles of induction chemotherapy (IC; gemcitabine-cisplatin regimen) followed by intensity-modulated radiotherapy (IMRT) alone. Nivolumab injection OPDIVO® will start on day 1 of the first cycle IC and continue every 3 weeks for 6 cycles till the end of IMRT, involving the whole-course of IC + IMRT alone. The first and last 3 cycles of nivolumab are administrated concurrently with IC and IMRT, respectively. After the completion of IMRT, adjuvant nivolumab will begin every 4 weeks for 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65;
2. Pathological type: non-keratinizing carcinoma (World Health Organization criteria);
3. Diagnosed with LANPC (T4N1, T1-4N2-3) according to the 8th edition clinical staging system of the American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC];
4. ECOG performance score: 0 to 1;
5. Normal bone marrow function: white blood cell count > 4×109/L, hemoglobin > 90g/L, platelet count > 100×109/L;
6. Normal values of thyroid function, amylase and lipase examination, pituitary function, inflammation and infection indicators, myocardial enzymes, and ECG results. For patients older than 50 years with a smoking history, normal lung function are required. Patients with abnormal ECG and/or a history of vascular disease (but not meeting the exclusion criteria listed in the exclusion criteria 7) need further testing and require normal results of myocardial function and color Doppler ultrasound.
7. Normal liver and kidney function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); alanine transaminase and aspartate transaminase ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; creatinine clearance rate ≥ 60 ml/min;
8. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;
9. Subjects with pregnancy ability must agree to use reliable contraceptive measures from screening to 1 year after treatment.

Exclusion Criteria:

1. Hepatitis B virus surface antigen (HBsAg) positive and HBV DNA > 1×10E3 copies/ml; anti-hepatitis C virus positive;
2. Anti-human immunodeficiency virus (HIV) positive or diagnosed with acquired immune deficiency syndrome (AIDS);
3. Active tuberculosis: active tuberculosis in the past 1 year should be excluded regardless with treatment; history of active tuberculosis over 1 year should be excluded except that previous regulatory anti-tuberculosis treatment is proved;
4. Active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchiectasis). Exceptions are type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia);
5. Previous interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy;
6. Chronic treatment with systemic glucocorticoid (dose equivalent to or over 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects who used inhaled or topical corticosteroids were eligible;
7. Uncontrolled heart disease, for example: 1) heart failure (NYHA level ≥ 2); 2) unstable angina; 3) myocardial infarction in past 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. Pregnant or lactating women (pregnancy test should be considered for women with sexual life and fertility);
9. Previous or concurrent with other malignant tumors, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary cancer;
10. Allergy to macromolecular protein preparations, or any component of nivolumab;
11. Active infection requiring systemic treatment;
12. Receiving live vaccine within 30 days of the initial nivolumab;
13. History of organ transplantation;
14. History of psychotropic disease, alcoholism or drug abuse; other situation assessed by the investigators that may compromise the safety or compliance of patients, such as serious disease requiring timely treatment (including mental illness), severe laboratory abnormalities, or family-social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3-year
  Failure-free survival is measured from day of enrollment until the first indication of treatment failure (either locoregional recurrence or distant metastasis) or death from any cause, whichever occurred first

SECONDARY OUTCOMES:
Overall survival (OS) | 3-year
  Overall survival is measured from day of enrollment until death due to any cause or the latest known date alive
Locoregional failure-free survival (LRFFS) | 3-year
  Locoregional failure-free survival is measured from day of enrollment until local or regional recurrence
Distant failure-free survival (DFFS) | 3-year
  Distant failure-free survival is measured from day of enrollment until distant metastasis
Incidence rate of investigator-reported adverse events (AEs) | 3-year
  Analysis of investigator-reported adverse events (AEs) are based on treatment-related AEs (trAEs) and immune-related AEs (irAEs), and all-grade AEs and grade 3-4 AEs. AEs are evaluated by investigators according to the Common Terminology Criteria for Adverse Events, version 5.0
Incidence rate of patient-reported adverse events (AEs) | 3-year
  Analysis of patient-reported adverse events (AEs) are based on the PRO-CTCAE. Tolerability profiles are evaluated by patients themselves.
Quality of life (QoL): questionnaire | baseline, week 7, 14, 38, 62
  Changes in QoL of participants from initial treatment to 6 months after the completion of 6 cycles adjuvant PD-1 blocking antibody. QoL is evaluated with the use of (1) the head-and-neck-specific module (H&N35) of the Quality of Life Questionnaire-Core 30 module (QLQ-C30), which is established by European Organization for Research and Treatment of Cancer (EORTC) and (2) the general and head-and-neck-specific module of the evaluation tool developed by the Functional Assessment of Cancer Therapy (FACT). Scores for the module range of H&N35 QLQ-C30 from 0 to 100, with higher scores indicating better functioning or well-being or higher symptom burden (scales measuring symptom burden were reverse-scored to facilitate presentation)

OTHER OUTCOMES:
Correlation between pre-treatment PD-L1 expression level and FFS | 3-year
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Correlation between pre-treatment PD-L1 expression level and OS | 3-year
  Pre-treatment PD-L1 expression level of tumor cell is evaluated centrally by means of immunohistochemical testing. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Correlation between the percentage of tumor-infiltrating lymphocytes (TILs) and PFS | 3-year
  TILs are lymphoid cells (T cells) that infiltrate solid tumors (intra-tumoral TILs) and stroma (stromal TILs), which play an important role in the tumor microenvironment. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Correlation between the percentage of tumor-infiltrating lymphocytes (TILs) and OS | 3-year
  TILs are lymphoid cells (T cells) that infiltrate solid tumors (intra-tumoral TILs) and stroma (stromal TILs), which play an important role in the tumor microenvironment. This is a single assessment with only one unit of measure, since the correlation is aimed to be roughly categorized into positive and negative.
Evaluate failure-free survival in the subgroup of age at diagnosis (year) | 3-year
  Subgroup analysis
Evaluate failure-free survival in the subgroup of gender (male and female) | 3-year
  Subgroup analysis
Evaluate failure-free survival in the subgroup of plasma Epstein-Barr virus DNA level | 3-year
  Subgroup analysis
Evaluate failure-free survival in the subgroup of clinical stage | 3-year
  Subgroup analysis
Evaluate the regression of tumor and parotid glands during radiotherapy | From the first fraction of radiotherapy to the end of treatment
  Evaluate the anatomical (size, volume, and 3-dimensional axis) and dosimetric changes of primary tumor, lymph node, and parotid glands during 33-fractionation radiotherapy by using cone beam computed tomography
Failure-free survival 2 (FFS 2) | within 10 years
  The time from randomization to the second or subsequent disease progression after the initiation of new anticancer therapy, or death from any cause, whichever occurred first.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, M.D., Principal Investigator — Sun Yat-sen University
Locations (6):
- China (6):
  - Fujian Provinve Cancer Hospital, Fuzhou, Fujian Provinve
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hubei Province Cancer Hosiptal, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Zhejiang Province Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No
We currently have no plans to share individual participant data.

REFERENCES:
- [Background] Zhang L, Huang Y, Hong S, Yang Y, Yu G, Jia J, Peng P, Wu X, Lin Q, Xi X, Peng J, Xu M, Chen D, Lu X, Wang R, Cao X, Chen X, Lin Z, Xiong J, Lin Q, Xie C, Li Z, Pan J, Li J, Wu S, Lian Y, Yang Q, Zhao C. Gemcitabine plus cisplatin versus fluorouracil plus cisplatin in recurrent or metastatic nasopharyngeal carcinoma: a multicentre, randomised, open-label, phase 3 trial. Lancet. 2016 Oct 15;388(10054):1883-1892. doi: 10.1016/S0140-6736(16)31388-5. Epub 2016 Aug 23. PMID 27567279
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Ma Y, Fang W, Zhang Y, Yang Y, Hong S, Zhao Y, Tendolkar A, Chen L, Xu D, Sheng J, Zhao H, Zhang L. A Phase I/II Open-Label Study of Nivolumab in Previously Treated Advanced or Recurrent Nasopharyngeal Carcinoma and Other Solid Tumors. Oncologist. 2019 Jul;24(7):891-e431. doi: 10.1634/theoncologist.2019-0284. Epub 2019 May 2. PMID 31048330
- [Background] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Background] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Background] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452
- [Background] Xu C, Zhang S, Li WF, Chen L, Mao YP, Guo Y, Liu Q, Ma J, Tang LL. Selection and Validation of Induction Chemotherapy Beneficiaries Among Patients With T3N0, T3N1, T4N0 Nasopharyngeal Carcinoma Using Epstein-Barr Virus DNA: A Joint Analysis of Real-World and Clinical Trial Data. Front Oncol. 2019 Nov 29;9:1343. doi: 10.3389/fonc.2019.01343. eCollection 2019. PMID 31850226
- [Derived] Li XM, Zhang XM, Li JY, Jiang N, Chen L, Tang LL, Mao YP, Li WF, Zhou GQ, Li YQ, Liu N, Zhang Y, Ma J. The immune modulation effects of gemcitabine plus cisplatin induction chemotherapy in nasopharyngeal carcinoma. Cancer Med. 2022 Sep;11(18):3437-3444. doi: 10.1002/cam4.4705. Epub 2022 Mar 30. PMID 35355438